CLINICAL TRIAL: NCT03652818
Title: Randomized, Double-blind, Parallel Group, Single-center, Placebo-controlled Study to Evaluate Efficacy and Safety of Analgesic Combo in Prevention and Treatment of Post-surgical Dental Pain in Healthy Subjects
Brief Title: Dental Pain Study of Analgesics in Patients Undergoing Molar Removal
Acronym: NVK009-0001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nevakar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP-NVK009-0001
Record Dates: First submitted 2018-07-18; First posted 2018-08-29 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The sponsor, patients, investigators and study staff involved in the protocol procedures or those involved in data collection, data entry, data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental): Pre-op Placebo 1;
  Post-op Placebo 1;
  Post-op Placebo 2
  Interventions: Drug: Pre-Op Placebo 1; Drug: Post-Op Placebo 1; Drug: Post-Op Placebo 2
- Group B (Experimental): Pre-op Placebo 1;
  Post-op Placebo 2;
  Post-op acetaminophen.
  Interventions: Drug: Pre-Op Placebo 1; Drug: Post-Op Placebo 1; Drug: Post-Op acetaminophen
- Group C (Experimental): Pre-op Placebo 1;
  Post-op pregabalin;
  Post-op Placebo 2.
  Interventions: Drug: Pre-Op Placebo 1; Drug: Post-Op pregabalin; Drug: Post-Op Placebo 2
- Group D (Experimental): Pre-op Placebo 1;
  Post-op pregabalin
  Post-op acetaminophen.
  Interventions: Drug: Pre-Op Placebo 1; Drug: Post-Op pregabalin; Drug: Post-Op acetaminophen
- Group E (Experimental): Pre-op pregabalin;
  Post-op Placebo 1;
  Post-op acetaminophen.
  Interventions: Drug: Pre-Op pregabalin; Drug: Post-Op Placebo 1; Drug: Post-Op acetaminophen

INTERVENTIONS:
Drug: Pre-Op pregabalin — Pre-op pregabalin will be administered 60 min prior to surgery.
  Arms: Group E
Drug: Pre-Op Placebo 1 — Placebo 1 will be administered 60 min prior to surgery.
  Other Names: pre-op placebo
  Arms: Group A; Group B; Group C; Group D
Drug: Post-Op pregabalin — Post-op pregabalin will be administered Post-operatively.
  Arms: Group C; Group D
Drug: Post-Op Placebo 1 — Placebo 1 will be administered post-operatively.
  Arms: Group A; Group B; Group E
Drug: Post-Op Placebo 2 — Placebo 2 will be administered post-operatively.
  Arms: Group A; Group C
Drug: Post-Op acetaminophen — Acetaminophen will be administered Post-operatively.
  Arms: Group B; Group D; Group E

SUMMARY:
* Accessing the efficacy and safety of pregabalin when used alone and in combo with acetaminophen in a dental pain model.
* To test whether pre-operative dose of pregabalin increases the time to significant post-operative pain (NRS ≥ 5), and hence time to first analgesia consumed post-operatively.

DETAILED DESCRIPTION:
This is a 5 arm randomized, double-blind, parallel group, single-center, placebo-controlled study to evaluate the efficacy and safety of pregabalin-acetaminophen combination in the prevention and treatment of post-surgical dental pain in healthy patients.

Subjects in every treatment arm will receive a dose 60 min prior to surgery. It is not required to receive a post-operative dose if patient does not feel pain at a scale of NRS≥ 5. Dose 2 will be given post-surgically when patients report at least moderate pain on the categorical scale and a score of ≥5 on 0-10 PI-NRS. Subsequent to dose 2, patients can request rescue analgesic at any time.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo the surgical removal of up to 4 third molars of which at least 2 have to be mandibular molars with a difficulty rating of 4 or 5.
* Patient must have a negative urine drug screen for drugs of abuse (including tobacco) at screening and at the day of surgery.
* No alcohol for a minimum of 1 day prior to the surgery.

Exclusion Criteria:

* Patients should not be experiencing oral infections or symptoms of concomitant illness at the time of a scheduled surgery.
* Patients with a history of any type of malignancy within the past 5 years other than minor skin related cancers.
* Patients who currently have or have had a history of uncontrolled hypertension.
* Patients with a known allergy or hypersensitivity to any local anesthetic drug, NSAIDs, gabapentin or pregabalin;.
* Patients with conditions that affect the absorption, metabolism, or passage of drugs out of the body (e.g., sprue, celiac disease, crohn's disease, etc.)

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Somberg, MD, Study Director — Nevakar, Inc.
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from June 2018 till September 2018 from the site
Pre-assignment Details: Participants were screened from Day-30 to Day 0 before getting randomized
Groups:
- Group A/ Placebo Group: Participants received matching placebo capsule orally 60 ± 10 minutes (min) prior to initiating the surgical procedure. Post-surgically the participants received matching placebo capsule orally and matching placebo (saline 100mL) intravenously (IV). The IV infusion was administered over a 15 min period and the capsule was administered immediately prior to the initiation of the IV infusion
- Group B/ Acetaminophen (APAP) 1000 mg IV Group: Participants received matching placebo capsule orally 60 ± 10 mins prior to initiating the surgical procedure. Post-surgically the participants received matching placebo capsule orally and APAP 1000 milligram (mg) IV. The IV infusion was administered over a 15 min period and the capsule was administered immediately prior to the initiation of the IV infusion.
- Group C/ Pregabalin (PGB) 300 mg Capsule Group: Participants received matching placebo capsule orally 60 ± 10 mins prior to initiating the surgical procedure. Post-surgically the participants received PGB 300 mg capsule orally and matching placebo (saline 100mL) IV. The IV infusion was administered over a 15 min period and the capsule was administered immediately prior to the initiation of the IV infusion.
- Group D/ Combination Co-dosing Group (Post-surgery PGB +APAP): Participants received matching placebo capsule orally 60 ± 10 mins prior to initiating the surgical procedure. Post-surgically the participants received PGB 300 mg capsule orally and APAP 100 mg IV. The IV infusion was administered over a 15 min period and the capsule was administered immediately prior to the initiation of the IV infusion.
- Group E/ Combination Split-dosing Group (PGB Pre-surgery + APAP Post-surgery): Participants received PGB 300 mg capsule orally 60 ± 10 mins prior to initiating the surgical procedure. Post-surgically the participants received matching placebo capsule orally and APAP 1000 mg IV. The IV infusion was administered over a 15 min period and the capsule was administered immediately prior to the initiation of the IV infusion
Period: Overall Study
Arm/Group | Group A/ Placebo Group | Group B/ Acetaminophen (APAP) 1000 mg IV Group | Group C/ Pregabalin (PGB) 300 mg Capsule Group | Group D/ Combination Co-dosing Group (Post-surgery PGB +APAP) | Group E/ Combination Split-dosing Group (PGB Pre-surgery + APAP Post-surgery)
Started | 24 | 23 | 22 | 23 | 23
Completed | 22 | 22 | 20 | 22 | 22
Not Completed | 2 | 1 | 2 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was randomized population, that included all randomized participants
Groups:
- Group A/ Placebo Group: Pre-surgery placebo and post-surgery placebo 1 and placebo 2
- Group B/ APAP Group: Pre-surgery placebo 1 and post-surgery placebo 1 and acetaminophen (APAP)
- Group C/ PGB Group: Pre-surgery placebo 1 and post-surgery placebo 2 and pregabalin (PGB)
- Group D/ Combination Co-dosing Group: Pre-surgery placebo 1 and post-surgery APAP and PGB
- Group E/ Combination Split-dosing Group: Pre-surgery PGB and post-surgery placebo 1 and APAP
- Total: Total of all reporting groups
Arm/Group | Group A/ Placebo Group | Group B/ APAP Group | Group C/ PGB Group | Group D/ Combination Co-dosing Group | Group E/ Combination Split-dosing Group | Total
Number analyzed (Participants) | 24 | 23 | 22 | 23 | 23 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.8 (1.79) | 17.8 (1.48) | 17.9 (1.39) | 17.7 (0.93) | 17.6 (1.31) | 17.7 (1.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 11 | 12 | 11 | 57
  Male | 12 | 12 | 11 | 11 | 12 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 4 | 2 | 9
  Not Hispanic or Latino | 23 | 21 | 22 | 19 | 21 | 106
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 22 | 21 | 22 | 22 | 23 | 110
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.86 (3.716) | 22.54 (3.227) | 22.78 (3.825) | 24.02 (3.788) | 23.85 (3.695) | 23.21 (3.642)
Number of Participants With Mandibular Molar - 17 [Count of Participants; unit: Participants] — Population: One participant from Placebo group (Group A) was withdrawn by physician prior to surgery due to emesis hence Baseline (Day 1) oral examinations was not conducted for this participant.
  Participants
    Moderate to severe partial bony: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Moderate to severe partial bony | 2 | 7 | 4 | 5 | 4 | 22
    Full bony impaction: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Full bony impaction | 21 | 16 | 18 | 18 | 19 | 92
Number of Participants With Mandibular Molar - 32 [Count of Participants; unit: Participants] — Population: One participant from Placebo group (Group A) was withdrawn by physician prior to surgery due to emesis hence Baseline (Day 1) oral examinations was not conducted for this participant.
  Participants
    Moderate to severe partial bony: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Moderate to severe partial bony | 4 | 7 | 5 | 4 | 3 | 23
    Full bony impaction: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Full bony impaction | 19 | 16 | 17 | 19 | 19 | 90
Number of Participants With Maxillary Molar -1 [Count of Participants; unit: Participants] — Population: One participant from Placebo group (Group A) was withdrawn by physician prior to surgery due to emesis hence Baseline (Day 1) oral examinations was not conducted for this participant.
  Participants
    Erupted in tissue: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Erupted in tissue | 2 | 1 | 1 | 0 | 0 | 4
    Soft tissue impaction: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Soft tissue impaction | 1 | 0 | 0 | 0 | 1 | 2
    Moderate to severe partial bony: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Moderate to severe partial bony | 0 | 2 | 3 | 2 | 0 | 7
    Full bony impaction: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Full bony impaction | 20 | 17 | 17 | 21 | 22 | 97
Number of Participants With Maxillary Molar -16 [Count of Participants; unit: Participants] — Population: One participant from Placebo group (Group A) was withdrawn by physician prior to surgery due to emesis hence Baseline (Day 1) oral examinations was not conducted for this participant.
  Participants
    Erupted in tissue: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Erupted in tissue | 0 | 0 | 0 | 1 | 0 | 1
    Soft tissue impaction: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Soft tissue impaction | 0 | 0 | 0 | 1 | 1 | 2
    Mild partial bony impaction: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Mild partial bony impaction | 0 | 0 | 1 | 0 | 0 | 1
    Moderate to severe partial bony: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Moderate to severe partial bony | 1 | 2 | 4 | 1 | 1 | 9
    Full bony impaction: number analyzed (Participants) | 23 | 23 | 22 | 23 | 23 | 114
    Full bony impaction | 22 | 19 | 15 | 20 | 21 | 97

OUTCOME MEASURES:

1. Primary Outcome: Sum Pain Intensity Difference Scores
Description: Beginning post-surgery (at initiation of Dose 2), Pain Intensity was self-reported over 24 hours, using a pain rating of 0-10 on the Numerical Rating Scale (NRS), with score between 0-10 (0= no pain; 10 = pain as bad as can be). Time weighted sum pain intensity difference scores are reported over 0 to 24 hours. Last observation carried forward method was used.
Time Frame: 0.5, 0.75, 1, 1.25, 1.75, 2.25 hours (± 5 min) and 3.25, 4.25, 5.25, 6.25, 8.25, 10.25, 12.25, 24 hours (± 10 min)
Population: Efficacy Analysis Population included all randomized participants who received study medication post-surgically and did not experience emesis or other major protocol deviations
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Group A/ Placebo Group | Group B/ APAP Group | Group C/ PGB Group | Group D/ Combination Co-dosing Group | Group E/ Combination Split-dosing Group
Number analyzed (Participants) | 19 | 23 | 21 | 22 | 10
score on a scale | -2.4292 (12.4980) | -68.0778 (11.2879) | -68.3533 (11.8092) | -93.3645 (11.5794) | -82.4099 (17.4418)
Statistical Analysis 1: Comparison: Group B/ APAP Group vs Group D/ Combination Co-dosing Group; Group D vs. Group B; Test type: Superiority; Least Square (LS) Mean Difference = -25.2868, 90% CI 1-sided [upper limit -4.4210], Standard Error of Mean 16.1594 — Statistics are from ANCOVA including treatment and sex as fixed effects with baseline PI score prior to Dose 2 as a covariate. The lower limit of one-sided 90% CI was -∞
Statistical Analysis 2: Comparison: Group B/ APAP Group vs Group C/ PGB Group; Group C vs. Group B; Test type: Superiority; LS Mean Difference = -0.2756, 90% CI 1-sided [upper limit 20.8083], Standard Error of Mean 16.3283 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group A/ Placebo Group vs Group C/ PGB Group; Group C vs. Group A; Test type: Superiority; LS Mean Difference = -65.9241, 90% CI 1-sided [upper limit -43.6959], Standard Error of Mean 17.2146 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group A/ Placebo Group vs Group B/ APAP Group; Group B vs. Group A; Test type: Superiority; LS Mean Difference = -65.6486, 90% CI 1-sided [upper limit -43.8584], Standard Error of Mean 16.8753 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group A/ Placebo Group vs Group D/ Combination Co-dosing Group; Group D vs. Group A; Test type: Superiority; LS Mean Difference = -90.9353, 90% CI 1-sided [upper limit -68.8494], Standard Error of Mean 17.1044 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group C/ PGB Group vs Group D/ Combination Co-dosing Group; Group D vs. Group C; Test type: Superiority; LS Mean Difference = -25.0112, 90% CI 1-sided [upper limit -3.6571], Standard Error of Mean 16.5376 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group D/ Combination Co-dosing Group vs Group E/ Combination Split-dosing Group; Group E vs. Group D; Test type: Superiority; LS Mean Difference = 10.9546, 90% CI 1-sided [upper limit 38.1014], Standard Error of Mean 21.0237 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Total Pain Relief Measure
Description: Beginning post-surgery (at initiation of Dose 2), Pain Relief was self-reported over 24 hours, using a pain rating of 0-10 on the Numerical Rating Scale (NRS), with score between 0-10 (0= no pain; 10 = pain as bad as can be). Time-weighted sum pain total pain relief scores over 24 hours is reported Last observation carried forward method was used.
Time Frame: 0.5, 0.75, 1, 1.25, 1.75, 2.25 hours (± 5 min) and 3.25, 4.25, 5.25, 6.25, 8.25, 10.25, 12.25, 24 hours (± 10 min)
Population: Efficacy Analysis Population: Included all randomized participants who received study medication post-surgically and did not experience emesis or other major protocol deviations
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Group A/ Placebo Group | Group B/ APAP Group | Group C/ PGB Group | Group D/ Combination Co-dosing Group | Group E/ Combination Split-dosing Group
Number analyzed (Participants) | 19 | 23 | 21 | 22 | 10
score on a scale | 17.1038 (15.5619) | 88.2775 (14.0551) | 94.4433 (14.7042) | 121.9596 (14.4180) | 91.8373 (21.7176)
Statistical Analysis 1: Comparison: Group B/ APAP Group vs Group D/ Combination Co-dosing Group; Group D vs. Group B; Test type: Superiority; LS Mean Difference = 33.6821, 90% CI 1-sided [lower limit 7.7011], Standard Error of Mean 20.1209 — Statistics are from ANCOVA including treatment and sex as fixed effects with baseline PI score prior to Dose 2 as a covariate. The upper limit was ∞
Statistical Analysis 2: Comparison: Group B/ APAP Group vs Group C/ PGB Group; Group C vs. Group B; Test type: Superiority; LS Mean Difference = 6.1658, 90% CI 1-sided [lower limit -20.0868], Standard Error of Mean 20.3312 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Group A/ Placebo Group vs Group C/ PGB Group; Group C vs. Group A; Test type: Superiority; LS Mean Difference = 77.3395, 90% CI 1-sided [lower limit 49.6620], Standard Error of Mean 21.4347 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Group A/ Placebo Group vs Group B/ APAP Group; Group B vs. Group A; Test type: Superiority; LS Mean Difference = 71.1737, 90% CI 1-sided [lower limit 44.0417], Standard Error of Mean 21.0123 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Group A/ Placebo Group vs Group D/ Combination Co-dosing Group; Group D vs. Group A; Test type: Superiority; LS Mean Difference = 104.8558, 90% CI 1-sided [lower limit 77.3555], Standard Error of Mean 21.2975 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Group C/ PGB Group vs Group D/ Combination Co-dosing Group; Group D vs. Group C; Test type: Superiority; LS Mean Difference = 27.5163, 90% CI 1-sided [lower limit 0.9272], Standard Error of Mean 20.5918 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Group D/ Combination Co-dosing Group vs Group E/ Combination Split-dosing Group; Group E vs. Group D; Test type: Superiority; LS Mean Difference = -30.1223, 90% CI 1-sided [lower limit -63.9240], Standard Error of Mean 26.1776 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Participants With Differing Patient Global Evaluation Scores
Description: Patient global evaluation was self-reported at time of first rescue or at 12.25 hours post-surgery, whichever was first, using a 0-4 categorical rating scale of: (0) poor, (1) fair, (2) good, (3) very good, and (4) excellent. The number of participants with differing patient global evaluation scores were reported.
Time Frame: Upto 12.25 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group A/ Placebo Group | Group B/ APAP Group | Group C/ PGB Group | Group D/ Combination Co-dosing Group | Group E/ Combination Split-dosing Group
Number analyzed (Participants) | 19 | 23 | 21 | 22 | 10
Participants
  (0) Poor | 13 | 1 | 8 | 0 | 0
  (1) Fair | 3 | 2 | 2 | 3 | 1
  (2) Good | 1 | 7 | 4 | 4 | 1
  (3) Very good | 2 | 8 | 6 | 10 | 6
  (4) Excellent | 0 | 5 | 1 | 5 | 2

4. Secondary Outcome: Cumulative Number of Participants With Onset of First Perceptible Relief (FPR) Confirmed at 24 Hours After Dose 2
Description: Beginning post-surgery (at initiation of Dose 2), participants were given a stopwatch and asked to press the stopwatch if and when they feel first perceptible relief; a record of the time was noted in the participants record. Cumulative number of participants with onset of FPR confirmed after dose 2 and was recorded from 0.25 hour till 24 hours after administration of dose 2.
Time Frame: 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0 and 24 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group A/ Placebo Group | Group B/ APAP Group | Group C/ PGB Group | Group D/ Combination Co-dosing Group | Group E/ Combination Split-dosing Group
Number analyzed (Participants) | 19 | 23 | 21 | 22 | 10
Participants | 12 | 23 | 17 | 22 | 10

5. Secondary Outcome: Cumulative Number of Participants With Onset of Meaning Pain Relief (MPR) Confirmed at 24 Hours After Dose 2
Description: Beginning post-surgery (at initiation of Dose 2), participants were given a stopwatch and asked to press the stopwatch if and when they feel first perceptible relief; a record of the time was noted in the participants record. Cumulative number of participants with onset of MPR confirmed after dose 2 and was recorded from 0.25 hour till 24 hours after administration of dose 2.
Time Frame: 0.25, 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0 and 24 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group A/ Placebo Group | Group B/ APAP Group | Group C/ PGB Group | Group D/ Combination Co-dosing Group | Group E/ Combination Split-dosing Group
Number analyzed (Participants) | 19 | 23 | 21 | 22 | 10
Participants | 3 | 20 | 11 | 17 | 10

ADVERSE EVENTS:
Time Frame: Up to Day 15 (± 1 day)
Description: An adverse event (AE) is defined as any untoward medical occurrence and does not necessarily have to have causal relationship with the study medication. An AE can therefore be an unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease, which is a change from baseline and is temporally associated with the use of the study medication, whether or not it is considered related to the study medication.
Arm/Group | Group A/ Placebo Group | Group B/ APAP Group | Group C/ PGB Group | Group D/ Combination Co-dosing Group | Group E/ Combination Split-dosing Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/22 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/22 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 2/24 | 3/23 | 14/22 | 15/23 | 12/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A/ Placebo Group (N=24) | Group B/ APAP Group (N=23) | Group C/ PGB Group (N=22) | Group D/ Combination Co-dosing Group (N=23) | Group E/ Combination Split-dosing Group (N=23)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 5 (5)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 9 (9) | 10 (10) | 3 (3)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 6 (6) | 6 (6) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT03652818/Prot_SAP_000.pdf